CLINICAL TRIAL: NCT01301651
Title: Effects of Virtual Reality Augmented Balance Training for Postural Control in Patients With Parkinson's Disease
Brief Title: Effects of Virtual Reality Training in Patients With Parkinson's Disease
Acronym: Parkinson
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 200712039R
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: Virtual Reality; Balance; Parkinson's disease; Dual Task
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- virtual reality balance training (Experimental): balance board training with virtual reality intervention
  Interventions: Behavioral: balance training
- conventional balance training (Experimental): physical therapy conventional balance training
  Interventions: Behavioral: balance training
- control group (No Intervention): No physical therapy

INTERVENTIONS:
Behavioral: balance training — 30 minute each time, 2 times per week for 6 weeks.
  Other Names: virtual reality
  Arms: conventional balance training; virtual reality balance training

SUMMARY:
Background and Objective: Postural instability is common in patient with Parkinson's disease (PD). The purpose of this study was to investigate the effects of virtual reality (VR) balance training on sensory and cognitive domains of postural control.

Setting: Balance Performance Laboratory. Participants: A total of 42 patients (Hoehn and Yahr stage II-III) were recruited and assigned into three groups randomly.

Intervention: Participants in the virtual reality (VR) group and conventional balance training (CB) group received a 6 weeks balance training program. The control group (CG) did not receive any training.

Outcome Measures: The sensory organization tests (SOT) of computerized dynamic posturography with single and dual tasks (i.e. with backward subtraction of number) were examined pre-, post-training and follow-up. The equilibrium score (ES) and sensory ratio were measured. The verbal reaction time (VRT) was recorded.

Results: (1) Only VR significantly increased ES of SOT-6 (i.e., vestibular function at visual and somatosensory conflicting condition) post-training more than CG post-training in either single or dual task. (2) Only CB training significantly increased SOT-5 (i.e., vestibular function without visual conflict) and vestibular sensory ratio (i.e., SOT-5/SOT-1) more than CG post-training in either single or dual task. (3) (3) Neither VR nor CB training reduced VRT significantly under six sensory conditions at post-training and follow-up.

Conclusion: Both VR training and CB training can improve sensory organization for postural control by enhancing utilization of vestibular information, but VR could enhance vestibular function with conflicting proprioceptive and visual information under single and dual tasks in patients with mild to moderate PD.

DETAILED DESCRIPTION:
It is common that people who are diagnosed with idiopathic Parkinson disease (PD) experience postural instability during daily activities.Recently, postural instability is suggested as the underlying mechanism of falling in patients with PD. Therefore, how to improve postural stability by balance training is an important issue for these patients.

Basal ganglia have been regarded to be predominantly involved in postural control. Several studies suggested that the dysfunction of basal ganglia in patients with PD might play a major role in postural instability. Furthermore, patients with PD might have impaired utilization of sensory information by the basal ganglia.Computerized dynamic posturography (CDP) has the Sensory Organization Test (SOT), which provides an objective assessment of the main sensory systems (i.e., vision, proprioception and vestibular system) involved in balance and stability. The role of sensory information under six conditions (i.e., eyes open, eyes closed, sway vision, eyes open sway support, eyes closed sway support, and sway vision sway support) has been studied in patients with PD by the SOT of computerized CDP. Their study indicated that patients with PD demonstrated a significant reduction in sensory integration of proprioception and vision, but no significant difference in vestibular function, as compared to age-matched controls. One study showed that patients with PD had visual dependence as an adaptive strategy partly compensating for the impaired proprioception. However, the other study suggested that the cerebellum might be important for sensory integration in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

(1) idiopathic Parkinson's disease, (2) intact cognition (Mini-Mental State Examination; MMSE>24), 22 (3) Hoehn and Yahr (H-Y) stage II-III diagnosed by neurologists, (4) not participated in any balance or gait training previously, (5) able to follow simple command and had no uncontrolled chronic condition.-

Exclusion Criteria:

(1) history of other neurological, cardiovascular and orthopedic diseases affecting postural stability, (2) on-off motor fluctuation and dyskinesia above grade 3 by the Unified Parkinson' Disease Scale (UPDRS)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The equilibrium score (ES) and sensory ratio were measured. The verbal reaction time (VRT) was recorded. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Hwa Lin, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Yen CY, Lin KH, Hu MH, Wu RM, Lu TW, Lin CH. Effects of virtual reality-augmented balance training on sensory organization and attentional demand for postural control in people with Parkinson disease: a randomized controlled trial. Phys Ther. 2011 Jun;91(6):862-74. doi: 10.2522/ptj.20100050. Epub 2011 Apr 7. PMID 21474638